CLINICAL TRIAL: NCT02757079
Title: Phase III Clinical Trial of NPC-15 - Study of the Efficacy and Safety for Sleep Disorders of Children With Neurodevelopmental Disorders -
Brief Title: Study of the Efficacy and Safety of NPC-15 for Sleep Disorders of Children With Neurodevelopmental Disorders
Acronym: NPC-15-6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-15-6
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorders; Neurodevelopmental Disorder
Keywords: Melatonin; NPC-15; Sleep disorders; Neurodevelopmental disorder; Sleep latency; DSM-5
MeSH Terms: conditions — Sleep Wake Disorders; Neurodevelopmental Disorders | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NPC-15 Granule (Experimental): NPC-15 granule 1 mg, 2 mg or 4 mg once a day, administered orally before going to bed.
  Interventions: Drug: NPC-15

INTERVENTIONS:
Drug: NPC-15 — NPC-15, Melatonin granule 1 mg, 2 mg or 4 mg, once a day, is administered orally before going to bed for 26 weeks after a screening phase of 2 weeks with placebo administration.
  Other Names: Melatonin

SUMMARY:
The purpose of this study is to evaluate the efficacy on sleep latency with electronic sleep diaries and the safety of NPC-15.

DETAILED DESCRIPTION:
This study will be a multicenter and open label trial. The trial has three phases; the screening phase, treatment phase and post-treatment phase. The screening phase comprises a screening visit where subject's initial eligibility will be evaluated. During open label treatment phase, all patients will be administered NPC-15 1 mg, 2 mg or 4 mg on the basis of their doctors' judgements.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients aged 6 to 15 years.
* Patients with "neurodevelopmental disorder" diagnosed by using DSM-5.
* Patients with average of daily sleep latency persisted over 30 min and the condition is continuous over 3 months
* Patients who are out-patient, not hospitalized patient.
* Signed informed consent obtained from rearer(s)/parent(s)/guardian(s) of the patient, or signed IC or informed assent obtained from the patient themselves.

Exclusion Criteria:

* Patients with at least severity in either Conceptual area, or Social area, or Practical area of intellectual disability have judged more than " the most severe" by using DSM-5.
* Patients who took melatonin (including supplement) in history.
* Patients who had taken Ramelteon within 4 weeks before clinical study starts.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Sleep latency with electronic sleep diary at week 10. | 10 weeks
  Sleep latency is a common endpoint in sleep disorders. In addition, it has been used in a randomized clinical study of sleep disorders of children with neurodevelopmental disorders.

SECONDARY OUTCOMES:
Sleep latency with electronic sleep diary at week 26. | 26 weeks
  To assess the efficacy of this drug in detail
Abnormal behavior checklist Japanese version | Week 10, 26
  To assess effects of this drug on neurodevelopment disorders
Adverse events | 28 weeks
  To assess safety of this drug
Laboratory findings, vital sign | 28 weeks
  To assess safety of this drug
Electro cardiogram | 28 weeks
  To assess safety of this drug

CONTACTS AND LOCATIONS:
Overall Officials: Yushiro Yamashita, MD, PhD, Principal Investigator — The Department of Pediatrics and Child Health Kurume University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided